CLINICAL TRIAL: NCT03701139
Title: Phacoemulsification Combined With Posterior Capsulotomy in Cataract Complicated With Primary Posterior Capsule Opacification: a Randomized Controlled Trial
Brief Title: Posterior Capsulotomy in Cataract Complicated With Primary Posterior Capsule Opacification.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhi Liu, Clinical Professor,director of Zhongshan Ophthalmic Center, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018KYPJ103
Record Dates: First submitted 2018-10-02; First posted 2018-10-09 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Cataract; Posterior Capsule Opacification
Keywords: phacoemulsification; cataract; primary posterior capsule opacification; posterior capsulotomy; randomized controlled trial; Nd:YAG laser capsulotomy
MeSH Terms: conditions — Cataract | interventions — Posterior Capsulotomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- posterior capsulotomy (Experimental): Primary posterior capsulotomy will be performed to remove the primary posterior capsule opacification after posterior capsule polishing during phacoemulsification.
  Interventions: Procedure: posterior capsulotomy
- Nd:YAG laser capsulotomy (Active Comparator): Nd:YAG laser capsulotomy will be performed 1 month postoperative to remove the primary posterior capsule opacification.
  Interventions: Procedure: laser capsulotomy

INTERVENTIONS:
Procedure: posterior capsulotomy — After phacoemulsification with intraocular lens implantation, primary posterior capsulotomy will be performed to remove the primary posterior capsule opacification after posterior capsule polishing. A limited anterior vitrectomy will be performed if the anterior hyaloid surface is broken.
  Arms: posterior capsulotomy
Procedure: laser capsulotomy — A routine phacoemulsification with intraocular lens implantation is performed. Then the Nd:YAG laser capsulotomy will be performed 1 month postoperative to remove the primary posterior capsule opacification.
  Arms: Nd:YAG laser capsulotomy

SUMMARY:
This is a two-arm, parallel group, open-label, randomized controlled trial to compare the visual acuity, visual quality, operative complications and the satisfaction of patients between primary posterior capsulorhexis group and laser capsulotomy group of cataract patients combined with primary posterior capsular opacification (PPCO).

DETAILED DESCRIPTION:
Primary posterior capsular opacification (PPCO) refers to the posterior capsule opacification which cannot be removed by polishing or vacuuming during cataract surgery. The surgeon may have to decide on primary posterior capsulorhexis or early neodymium-doped yttrium aluminum garnet (Nd:YAG) laser capsulotomy in these cases. The aim of this study is to compare the visual acuity, visual quality, operative complications and the satisfaction of patients between primary posterior capsulorhexis group and laser capsulotomy group of cataract patients combined with primary posterior capsular opacification (PPCO).

ELIGIBILITY:
Inclusion Criteria:

1. Cataract patients with primary posterior capsular opacification, which involves the central posterior capsular and interferes with visual axis;
2. Aged 18 years or over;
3. With best corrected visual acuity (BCVA) less than 0.3.

Exclusion Criteria:

1. History of other eye disease that contributes to visual impairment, including keratopathy, uveitis, glaucoma, retinopathy, ocular trauma, or intraocular surgery.
2. Cases with operative complications, including anterior or posterior capsular rupture, lens suspensory ligament rupture, the falling of lens nucleus into vitreous cavity.
3. Unwillingness to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
LogMAR visual acuity 1 month postoperatively | 1 month
  Best corrected visual acuity (LogMAR) will be measured 1 month postoperatively.

SECONDARY OUTCOMES:
Dysfunctional lens index (DLI) | 3 months
  The dysfunctional lens index (DLI) is an objective lens performance metric derived from internal higher order aberrations (HOAs), pupil size, and contrast sensitivity data. DLI is a score ranged from 0 to 10. DLI will be measured by iTrace aberrometer.
Internal higher order aberration (HOAs) | 3 months
  TInternal higher order aberration (HOAs) in micrometer can quantify the intraocular optical quality and will be measured by iTrace aberrometer.
Object scatter index (OSI) | 3 months
  Object scatter index (OSI) is a ratio of 12 and 20 points from the perspective of the annular region of the light and the central 1 point perspective peak. OSI can objectively evaluate the amount of intraocular scattering and is an important index of optical quality. OSI is a score ranged from 0 to 10 and will be measured by Optical Quality Analysis System (OQAS).
Modulation transfer function cut off (MTF cut off) | 3 months
  Modulation transfer function cut off (MTF cut off) relates directly to retinal image quality and is a useful indicator of visual performance in cataract eyes. MTF cut off will be measured by OQAS.
Strehl ratio (SR) | 3 months
  Strehl ratio (SR) is computed as the ratio between the areas under the MTF curve of the measured eye and that of the aberration-free eye, and therefore it provides more global information on the optical quality. SR is a score ranged from 0 to 1 and will be measured by OQAS.
Predicted visual acuity (PVA) with contrasts of 100%, 20% and 10% | 3 months
  Predicted visual acuity (PVA) with contrasts of 100%, 20% and 10% correspond to three specific frequencies of the MTF that describe the eye's optical quality for the contrast values mentioned. In general, PVAs higher than 1 are associated to very high retinal image quality. PVA will be measured by OQAS.
Rate of ocular hypertension | 3 months
  Diagnosis of ocular hypertension is based on IOP greater than 21 mm Hg and the rate of ocular hypertension is calculated.
Rate of ocular macular edema | 3 months
  The central macular thickness in micrometer is measured by optical coherence tomography (OCT) and the rate of ocular macular edema is calculated.
Rate of retinal detachment | 3 months
  Retinal detachment following surgical or laser posterior capsulotomy is documented and the rate of Retinal detachment is calculated.
Rate of intraocular lens damage | 3 months
  The rate of intraocular lens damage by Nd:YAG laser is documented.
Visual-functioning index 7 score | 3 months
  Subjective satisfaction of patients is investigated by visual-functioning index 7 (VF-7) questionnaire. The VF-7 questionnaire comprises 7 questions for performing daily-life activities (1= a great deal of difficulty; 2= a moderate amount difficulty; 3= a little difficulty; 4= no difficulty). The VF-7 score is the average score of these 7 activities multiplied by 25, to give a final score between 0 and 100.
  1. nighttime driving;
  2. reading small print;
  3. watching television;
  4. seeing steps, stairs, or curbs;
  5. reading traffic, street, or store signs;
  6. cooking;
  7. doing fine handwork

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, PhD, Principal Investigator — Zhongshan Ophthamic Center,Sun Yet-san University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China